CLINICAL TRIAL: NCT00555724
Title: A Phase 1, Open Label, Dose Escalation Study of BIIB022 (Anti-IGF-1R Monoclonal Antibody) in Subjects With Relapsed or Refractory Solid Tumors
Brief Title: Phase 1 Study of BIIB022 (Anti-IGF-1R Monoclonal Antibody) in Relapsed/Refractory Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 212ST101
Record Dates: First submitted 2007-10-31; First posted 2007-11-09 (Estimated); Last update posted 2017-01-09 (Estimated); Status verified 2017-01

CONDITIONS: Solid Tumors
Keywords: Relapsed; refractory; solid tumor
MeSH Terms: conditions — Recurrence | interventions — BIIB022; Receptor Protein-Tyrosine Kinases

ARMS (1):
- BIIB022 (Experimental)
  Interventions: Drug: BIIB022

INTERVENTIONS:
Drug: BIIB022 — IV infusion once every three weeks until disease progression or unacceptable toxicity
  Other Names: IGF-1R

SUMMARY:
Phase 1, open-labeled, dose escalation safety and tolerability study for the treatment of subjects with relapsed or refractory solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older at the time of informed consent
* Relapsed or refractory solid tumors following standard therapy.
* ECOG Performance Status 0 or 1.

Exclusion Criteria:

* History of insulin-dependent diabetes, type 2 diabetes, or hemoglobin A1c >6% at screening.
* History of myocardial infarction within 12 months prior to Day 1 or chronic heart failure.
* Known central nervous system or brain metastases.
* Prior anti-IGF-1R therapy of any kind.

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-01; Primary Completion 2010-04 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of BIIB022 | ongoing

SECONDARY OUTCOMES:
To evaluate pharmacokinetics | ongoing

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Research Site, Los Angeles, California
  - Research Site, Aurora, Colorado
  - Research Site, Philadelphia, Pennsylvania

REFERENCES:
- [Background] von Mehren M, Britten CD, Pieslor P, Saville W, Vassos A, Harris S, Galluppi GR, Darif M, Wainberg ZA, Cohen RB, Leong S. A phase 1, open-label, dose-escalation study of BIIB022 (anti-IGF-1R monoclonal antibody) in subjects with relapsed or refractory solid tumors. Invest New Drugs. 2014 Jun;32(3):518-25. doi: 10.1007/s10637-014-0064-y. Epub 2014 Jan 24. PMID 24458261